CLINICAL TRIAL: NCT07386301
Title: Open Membrane Technique as an Innovative Minimally Invasive Technique for Hard and Soft Tissue Augmentation: a Retrospective Case Series
Brief Title: Open Membrane Technique as an Innovative Minimally Invasive Technique for Bone Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Abdel Rahman Kassir, Clinical Instructor, Saint-Joseph University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: USJ-2023 241
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Bone Graft; Keratinized Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients requiring horizontal bone augmentation in the posterior mandible (Other)
  Interventions: Procedure: Bone Augmentation

INTERVENTIONS:
Procedure: Bone Augmentation — Dense PTFE membranes covering an allograft biomaterial were used without any attempt to passivate the flap

SUMMARY:
Sixteen patients with horizontal deficiencies in the posterior mandible were treated with "the Open Membrane Technique" (OMT). Dense PTFE membranes covering an allograft biomaterial were used without any attempt to passivate the flap. Flap closure with an open wound (membrane exposure) was monitored weekly for up to 6w at the time of membrane removal. At implant placement, soft and hard tissue gains were assessed clinically and radiographically. Bone cores were harvested for histological analysis from the implant preparation sites

ELIGIBILITY:
Inclusion Criteria:

Healthy adults Free of any systemic disease affecting bone metabolism Highly compliant Good oral hygiene Willing to sign informed consents prior to their inclusion

Exclusion Criteria:

Untreated periodontal disease Heavy smokers Excessive alcohol consumption Uncontrolled systemic conditions

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Hard tissue gain | 5 months
  Bone thickness measured clinically and on CBCT (during bone grafting and at re-entry)

SECONDARY OUTCOMES:
Soft Tissue Gain | 5 months
  Keratinized tissue measured clinically before and after the treatment (at implant placement)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic 506, Beirut, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Any data will be shared with other researches if it is required or will help conducting further studies.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data are available at any time